CLINICAL TRIAL: NCT02851303
Title: Morphine Versus Methadone for Opiate Exposed Infants With Neonatal Abstinence Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Mary Beth Sutter, Attending Physician, Assistant Professor, University of New Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-176
Record Dates: First submitted 2016-07-19; First posted 2016-08-01 (Estimated); Results first posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Neonatal Abstinence Syndrome
MeSH Terms: conditions — Neonatal Abstinence Syndrome | interventions — Morphine; Methadone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Morphine (Active Comparator): Dose given q 3 - 4 hrs with feeds; do not exceed 4 hrs between doses Morphine (0.04mg/0.1ml)
  Score Dose For Initiation 0-8 0 None 9-12 0.04 mg/dose 13-16 0.08 mg/dose 17-20 0.12 mg/dose 21-24 0.16 mg/dose 25 or above 0.20mg/dose
  Morphine Maintenance/Escalation
  * Maintain dose if score 0-8
  * Increase dose by 0.02 if score is 9-12 (rescore before dosing) • Increase dose by 0.04 if score 13-16
  * Increase score by 0.06 if score 17-20
  Weaning Instructions:
  * Maintain on dose 48 hrs before starting weaning
  * Wean 0.02 mg morphine every day for a score is 0-8 • Defer wean for score 9-12
  Re-escalation
  * If neonate scores 9-12 re-score as described for initiation,
  * If second score is in 9-12 increase morphine 0.01 mg q3-4 hrs • If 2 consecutive scores 13-16, increase 0.02 mg q3-4 hrs
  * If 2 consecutive scores in 17-20, increase 0.04 mg q3-4 hrs etc
  Interventions: Drug: Morphine
- Methadone (Active Comparator): Step 1: 0.7 mgs/Kg/24 hrs. divided by into six doses (q 4 hrs) is starting dose Step 2: Decrease dose by half, which is 50% of starting dose, EVERY 4 hours. Step 3: Same dose which is 50% of starting dose EVERY 6 hours. Step 4: Same dose which is 50% of starting dose EVERY 8 hours. Step 5: Same dose which is 50% of starting dose EVERY 12 hours. Step 6: Decrease dose by half, which is 25% of starting dose EVERY 12 hours. Step 7: Same dose which is 25% of starting dose q 24 hours
  Interventions: Drug: Methadone

INTERVENTIONS:
Drug: Morphine — Morphine wean protocol as described in arm description
  Arms: Morphine
Drug: Methadone — Methadone wean protocol as described in arm description
  Arms: Methadone

SUMMARY:
This study investigates the use of methadone versus morphine wean for the treatment of neonatal abstinence syndrome for infants exposed to opioids in utero. Half of infants who require pharmacotherapy for NAS will receive a methadone wean, and half will receive a morphine wean. Length of hospital stay, length of treatment and parent satisfaction will be studied.

DETAILED DESCRIPTION:
Neonates exposed to opiates in utero can develop a constellation of withdrawal symptoms known as neonatal abstinence syndrome (NAS). Infants with NAS are at risk for multiple medical complications including failure to thrive and seizures, they often require prolonged hospital stays and account for significant health care costs. At University of New Mexico, infants exposed to methadone or heroin in utero who develop NAS requiring pharmacologic treatment undergo a treatment wean with methadone, whereas infants exposed to buprenorphine undergo a wean with morphine. However, morphine is used frequently to treat neonatal abstinence syndrome among methadone-exposed infants throughout the US, and optimal pharmacologic treatment for NAS remains unknown. Anecdotal evidence at the investigators institution suggests that infants treated with morphine have shorter hospital stays compared to infants treated with methadone. Investigators propose a pilot randomized controlled trial to evaluate morphine vs methadone treatment of infants with in-utero methadone or heroin exposure. Specifically, length of treatment, need for additional medication to treat withdrawal, and length of hospital stay will be compared.

When women are admitted to Labor and Delivery and/or up to 12 hours postpartum, research staff will approach patients about study enrollment. Participants will be approached for study enrollment if medication list on admission includes methadone, if participants self-report methadone use prenatally, and/ or if urine drug screen is positive for methadone or opiates on admission. If women choose to enroll in the study, and their infants require treatment for NAS, their infants will be randomized and assigned a study number for treatment using the methadone or morphine protocols at the time treatment is required.

All infants will be monitored for signs of withdrawal using the standard UNM NAS scoring protocol. Standard of care at UNM is to treat infants exposed to opioids in-utero with methadone if they require pharmacologic therapy for NAS, therefore treatment will not be withheld if they choose not to enroll in the study. Standard of care is also to obtain a urine drug screen on all infants with reported exposure to opiates in pregnancy. Enrolled patients will thus undergo routine urine drug screening. The only difference from standard care with regards to the study protocol is the treatment of half of the methadone or heroin exposed infants with morphine. The morphine protocol is proven for safety and efficacy currently in buprenorphine exposed infants. Once randomized, infants will continue on the protocol until discharge. At discharge, parents will complete a patient satisfaction survey.

ELIGIBILITY:
Inclusion criteria:

* Born at University of New Mexico Hospital
* Greater than 34 weeks gestation
* Primary in-utero drug exposure was opioids other than buprenorphine
* Maternal or infant urine drug screen positive for methadone and/or opioids on admission

Exclusion criteria:

* Born prior to 34 weeks
* Neonatal intensive care unit admission
* Serious medical comorbidities
* Primary substance exposure in-utero was buprenorphine, or was not opioids

Ages: 0 Hours to 12 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2016-10; Primary Completion 2018-06 (Actual); Study Completion 2018-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Beth Sutter, MD, Principal Investigator — Attending Physician, Assistant Professor
Locations (1):
- University of New Mexico Health Sciences Center, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hudak ML, Tan RC; COMMITTEE ON DRUGS; COMMITTEE ON FETUS AND NEWBORN; American Academy of Pediatrics. Neonatal drug withdrawal. Pediatrics. 2012 Feb;129(2):e540-60. doi: 10.1542/peds.2011-3212. Epub 2012 Jan 30. PMID 22291123
- [Background] Patrick SW, Davis MM, Lehmann CU, Cooper WO. Increasing incidence and geographic distribution of neonatal abstinence syndrome: United States 2009 to 2012. J Perinatol. 2015 Aug;35(8):650-5. doi: 10.1038/jp.2015.36. Epub 2015 Apr 30. PMID 25927272
- [Background] Hall ES, Wexelblatt SL, Crowley M, Grow JL, Jasin LR, Klebanoff MA, McClead RE, Meinzen-Derr J, Mohan VK, Stein H, Walsh MC; OCHNAS Consortium. A multicenter cohort study of treatments and hospital outcomes in neonatal abstinence syndrome. Pediatrics. 2014 Aug;134(2):e527-34. doi: 10.1542/peds.2013-4036. PMID 25070317
- [Background] Winter M, Nelson DS, Milton GW. Leucocyte adherence inhibition test for the detection of cell-mediated immunity to malignant melanoma. Aust N Z J Med. 1980 Aug;10(4):405-9. doi: 10.1111/j.1445-5994.1980.tb04090.x. PMID 7000060
- [Background] Logan BA, Brown MS, Hayes MJ. Neonatal abstinence syndrome: treatment and pediatric outcomes. Clin Obstet Gynecol. 2013 Mar;56(1):186-92. doi: 10.1097/GRF.0b013e31827feea4. PMID 23314720
- [Background] Hall ES, Wexelblatt SL, Crowley M, Grow JL, Jasin LR, Klebanoff MA, McClead RE, Meinzen-Derr J, Mohan VK, Stein H, Walsh MC; OCHNAS Consortium. Implementation of a Neonatal Abstinence Syndrome Weaning Protocol: A Multicenter Cohort Study. Pediatrics. 2015 Oct;136(4):e803-10. doi: 10.1542/peds.2015-1141. Epub 2015 Sep 14. PMID 26371196
- [Background] Jones HE, Kaltenbach K, Heil SH, Stine SM, Coyle MG, Arria AM, O'Grady KE, Selby P, Martin PR, Fischer G. Neonatal abstinence syndrome after methadone or buprenorphine exposure. N Engl J Med. 2010 Dec 9;363(24):2320-31. doi: 10.1056/NEJMoa1005359. PMID 21142534
- [Derived] Sutter MB, Watson H, Yonke N, Weitzen S, Leeman L. Morphine versus methadone for neonatal opioid withdrawal syndrome: a randomized controlled pilot study. BMC Pediatr. 2022 Jun 15;22(1):345. doi: 10.1186/s12887-022-03401-3. PMID 35705944
- [Derived] Zankl A, Martin J, Davey JG, Osborn DA. Opioid treatment for opioid withdrawal in newborn infants. Cochrane Database Syst Rev. 2021 Jul 7;7(7):CD002059. doi: 10.1002/14651858.CD002059.pub4. PMID 34231914

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were enrolled as dyads during the initial birth hospitalization. Randomization occured at the time of consent to allow for pharmacologic treatment to begin whenever it was deemed medically necessary without the time constraint of needing randomization by the research team. As not all infants required pharmacologic treatment for withdrawal, they dropped out of the study arm.
Groups:
- Morphine: Dose given q 3 - 4 hrs with feeds; do not exceed 4 hrs between doses Morphine (0.04mg/0.1ml)
  Score Dose For Initiation 0-8 0 None 9-12 0.04 mg/dose 13-16 0.08 mg/dose 17-20 0.12 mg/dose 21-24 0.16 mg/dose 25 or above 0.20mg/dose
  Morphine Maintenance/Escalation
  * Maintain dose if score 0-8
  * Increase dose by 0.02 if score is 9-12 (rescore before dosing) • Increase dose by 0.04 if score 13-16
  * Increase score by 0.06 if score 17-20
  Weaning Instructions:
  * Maintain on dose 48 hrs before starting weaning
  * Wean 0.02 mg morphine every day for a score is 0-8 • Defer wean for score 9-12
  Re-escalation
  * If neonate scores 9-12 re-score as described for initiation,
  * If second score is in 9-12 increase morphine 0.01 mg q3-4 hrs • If 2 consecutive scores 13-16, increase 0.02 mg q3-4 hrs
  * If 2 consecutive scores in 17-20, increase 0.04 mg q3-4 hrs etc
  Morphine: Morphine wean protocol as described in arm description
Period: Overall Study
Arm/Group | Morphine | Methadone
Started | 15 (Parent-Infant Dyads) | 13 (Parent-Infant Dyads)
Completed | 15 (Parent-Infant Dyads) | 13 (Parent-Infant Dyads)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 28 out of 61 randomized required pharmacologic therapy for withdrawal. Participant number reflects dyad pairs. Data collected from parent and or infant as described in footnotes for each item. Data were not collected for infants on items other than gestational age at birth.
Groups:
- Total: Total of all reporting groups
Arm/Group | Morphine | Methadone | Total
Number analyzed (Participants) | 15 | 13 | 28
Age, Continuous [Mean (Standard Deviation); unit: weeks] — Gestational age of infant component of the dyad at birth
  weeks | 37.7 (1.7) | 37.5 (1.2) | 37.6 (1.5)
Age, Customized [Mean (Standard Deviation); unit: years] — Age of parent component of the dyad
  years
    Mean age | 27.8 (4.3) | 25.4 (3.1) | 26.68 (3.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Reflects parent component of dyad
  Participants
    Female | 15 | 13 | 28
    Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Reflects parent component of dyad
  Participants
    White non-hispanic | 2 | 6 | 8
    hispanic | 11 | 7 | 18
    native american | 2 | 0 | 2
Initiation of prenatal care in first trimester [Count of Participants; unit: Participants] — Reflects parent component of dyad
  Participants | 5 | 9 | 14
Concurrent illicit opioid use [Count of Participants; unit: Participants] — Reflects parent component of dyad
  Participants | 12 | 10 | 22
Concurrent tobacco use [Count of Participants; unit: Participants] — Reflects parent component of dyad
  Participants | 9 | 6 | 15
Concurrent methamphetamine use [Count of Participants; unit: Participants] — Reflects parent component of dyad
  Participants | 10 | 2 | 12
Concurrent benzodiazepine use [Count of Participants; unit: Participants] — Reflects parent component of dyad
  Participants | 4 | 0 | 4
Concurrent alcohol use [Count of Participants; unit: Participants] — Reflects parent component of dyad
  Participants | 0 | 0 | 0
Concurrent SSRI [Count of Participants; unit: Participants] — Reflects parent component of dyad
  Participants | 2 | 0 | 2
Preterm delivery [Count of Participants; unit: Participants] — Reflects parent component of dyad/ birth gestational age of infant component of dyad
  Participants | 4 | 2 | 6
Maternal gestational diabetes [Count of Participants; unit: Participants] — Reflects parent component of dyad
  Participants | 1 | 0 | 1
Maternal preeclampsia [Count of Participants; unit: Participants] — Reflects parent component of dyad
  Participants | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Length of Hospital Stay
Description: Number of days in hospital after birth
Time Frame: assessed at hospital discharge, approximately 7-30 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Morphine | Methadone
Number analyzed (Participants) | 15 | 13
days | 17.9 (8.6) | 16.1 (4.7)

2. Secondary Outcome: Length of Treatment
Time Frame: assessed at hospital discharge, approximately 7-30 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Morphine | Methadone
Number analyzed (Participants) | 15 | 13
days | 14.7 (9.9) | 12.8 (5.8)

3. Secondary Outcome: Need for Additional Agent to Treat Withdrawal, Determined by Chart Review of Medication Administration Record of Administered Medications for Withdrawal Treatment (Example: Clonidine or Phenobarbital)
Description: clonidine
Time Frame: assessed at hospital discharge, approximately 7-30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Morphine | Methadone
Number analyzed (Participants) | 15 | 13
Participants | 1 | 0

4. Secondary Outcome: Need for Feeding Assistance, Determined by Chart Review of Discharge Summary, Specifically Evaluating for Need for Nasogastric Tube Placement or Peripheral Parenteral Nutrition.
Time Frame: assessed at hospital discharge, approximately 7-30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Morphine | Methadone
Number analyzed (Participants) | 15 | 13
Participants | 11 | 6

5. Secondary Outcome: Need for NICU Transfer, as Determined by Chart Review of Discharge Summary.
Time Frame: assessed at hospital discharge, approximately 7-30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Morphine | Methadone
Number analyzed (Participants) | 15 | 13
Participants | 0 | 3

6. Secondary Outcome: Breastfeeding Initiation and Continuation at Hospital Discharge
Description: Assessed through chart review of discharge summary documentation of method of infant feeding at time of discharge
Time Frame: assessed at hospital discharge, approximately 7-30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Morphine | Methadone
Number analyzed (Participants) | 15 | 13
Participants | 5 | 5

7. Secondary Outcome: Total Morphine Equivalent Dose Received
Time Frame: assessed at hospital discharge, approximately 7-30 days
Measure: Mean (Standard Deviation); unit: morphine equivalents mg
Arm/Group | Morphine | Methadone
Number analyzed (Participants) | 15 | 13
morphine equivalents mg | 9.86 (12.92) | 33.0 (17.49)

ADVERSE EVENTS:
Time Frame: Collected during initial hospitalization following birth for entire length of hospital stay on infants of dyads only. No infant adverse events following hospital discharge were collected. No maternal adverse events were examined/collected.
Groups:
- Morphine: Dose given q 3 - 4 hrs with feeds; do not exceed 4 hrs between doses Morphine (0.04mg/0.1ml)
  Score Dose For Initiation 0-8 0 None 9-12 0.04 mg/dose 13-16 0.08 mg/dose 17-20 0.12 mg/dose 21-24 0.16 mg/dose 25 or above 0.20mg/dose
  Morphine Maintenance/Escalation
  * Maintain dose if score 0-8
  * Increase dose by 0.02 if score is 9-12 (rescore before dosing) • Increase dose by 0.04 if score 13-16
  * Increase score by 0.06 if score 17-20
  Weaning Instructions:
  * Maintain on dose 48 hrs before starting weaning
  * Wean 0.02 mg morphine every day for a score is 0-8 • Defer wean for score 9-12
  Re-escalation
  * If neonate scores 9-12 re-score as described for initiation,
  * If second score is in 9-12 increase morphine 0.01 mg q3-4 hrs • If 2 consecutive scores 13-16, increase 0.02 mg q3-4 hrs
  * If 2 consecutive scores in 17-20, increase 0.04 mg q3-4 hrs etc
  Morphine: Morphine wean protocol as described in arm description
  Adverse events were recorded only for infants of each dyad.
- Methadone: Step 1: 0.7 mgs/Kg/24 hrs. divided by into six doses (q 4 hrs) is starting dose Step 2: Decrease dose by half, which is 50% of starting dose, EVERY 4 hours. Step 3: Same dose which is 50% of starting dose EVERY 6 hours. Step 4: Same dose which is 50% of starting dose EVERY 8 hours. Step 5: Same dose which is 50% of starting dose EVERY 12 hours. Step 6: Decrease dose by half, which is 25% of starting dose EVERY 12 hours. Step 7: Same dose which is 25% of starting dose q 24 hours
  Methadone: Methadone wean protocol as described in arm description
  Adverse events were recorded only for infants of each dyad.
Arm/Group | Morphine | Methadone
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/13
Other Adverse Events (participants affected / at risk) | 0/15 | 3/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Morphine (N=15) | Methadone (N=13)
High level of care transfer (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 3 (3) — Baby had to be transferred to higher level of care for over sedation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-04-09): https://cdn.clinicaltrials.gov/large-docs/03/NCT02851303/Prot_SAP_000.pdf
  • Informed Consent Form (2018-04-09): https://cdn.clinicaltrials.gov/large-docs/03/NCT02851303/ICF_001.pdf